CLINICAL TRIAL: NCT03134495
Title: A Cohort Study to Assess the Impact of Paediatric Use of Proton Pump Inhibitors on the Risk of Community Acquired Infections
Brief Title: the Impact of Paediatric Use of Proton Pump Inhibitors on the Risk of Community Acquired Infections.
Acronym: UTOPIE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LUU 2017
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Community Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PPI exposed children: all children with at least one prescription of PPI
  Interventions: Other: all children with at least one prescription of PPI
- non-exposed children: all children with no prescription of PPI
  Interventions: Other: all children with no prescription of PPI

INTERVENTIONS:
Other: all children with at least one prescription of PPI — all children with at least one prescription of PPI
  Groups: PPI exposed children
Other: all children with no prescription of PPI — all children with no prescription of PPI
  Groups: non-exposed children

SUMMARY:
Pharmacological treatment of physiologic Gastro-esophageal Reflux disease (GERD) is excessive in France, as 65%-85% of children below 11 years are being treated, frequently with Proton Pump Inhibitors (PPIs) PPI have been associated, in adults, with an increase of infection rate but data in pediatry are scarce, especially in community medecine. Recently a study conducted in England brought up controversial results suggesting that the use of PPIs can be associated with a reduced risk of community acquired pneumonia.

Our study was aimed to assess, on a population-based database, the association between PPI prescription and community infections in children of 11 years or under.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 11 years or below with at least 2 consultations during the follow up

Exclusion Criteria:

* chronic pulmonary or cardiac
* muscoviscidosis
* immunodeficiency
* H. pylori infection
* Diabetes
* Denutrition
* known digestive upper tract malformation

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all children included in the LDP-CSD database (Cegedim©) aged 11 or below, between 01/01/2008 and 31/12/2013
Sampling Method: Non-Probability Sample
Enrollment: 290286 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of overall infections | 4 years
  Comparison of number of infections between PPI exposed and non-exposed children. All infections are taken in account

SECONDARY OUTCOMES:
Number of specific infections | 4 years
  Comparison of number of infections between PPI exposed and non-exposed

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Dijon, Dijon, France